CLINICAL TRIAL: NCT01942837
Title: Phase II Trial of Enzalutamide for Castrate-resistant Prostate Cancer (CRPC) With Correlative Assessment of Androgen Receptor (AR) Signaling and Whole-exome and Transcriptome Sequencing
Brief Title: Study of Enzalutamide in Patients With Castration-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-301
Record Dates: First submitted 2013-09-04; First posted 2013-09-16 (Estimated); Results first posted 2022-07-05 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Enzalutamide; Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzalutamide (Experimental): Administration: 160 mg orally once daily with a 28-day cycle. Treatment will be continued until evidence of symptomatic or radiographic progression or the participant is taken off the study for another reason.
  Dosing: 160 mg orally taken once daily as four 40 mg capsules.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Enzalutamide, formerly known as MDV3100, is a rationally-designed second generation AR inhibitor which functions by blocking several steps in the AR signaling cascade. Enzalutamide competitively binds the AR with great potency. Additionally, enzalutamide inhibits nuclear translocation of activated AR and inhibits the association of activated AR with DNA.
  Other Names: Xtandi

SUMMARY:
This research study is evaluating a drug called enzalutamide in metastatic castration resistant prostate cancer. Enzalutamide is already FDA approved for metastatic castration resistant prostate cancer after treatment with chemotherapy.

The purpose of this study is to analyze features of tumor specimens sampled prior to therapy and at disease progression to determine why patients respond or stop responding to treatment with Enzalutamide.

Prior chemotherapy is not a requirement of this trial.

DETAILED DESCRIPTION:
After the screening procedures confirm that the patient is able to participate in the study,

* The patient will have the first of two required prostate biopsies prior to starting study treatment.
* The patient will be given a prescription for study drug and a study drug-dosing diary for each treatment cycle. Each treatment cycle lasts 28 days (4 weeks), during which time the patient will be taking the study drug once daily. The diary will also include special instructions for taking the study drug. The study drug (enzalutamide) should be taken orally (by mouth) at home.

On Day 1 of each cycle (+/- 4 days), the following procedures will be performed in clinic:

* A medical history.
* A Physical examination
* Performance status
* Blood tests (2-3 tablespoons).
* The patient will be asked about medications they are currently taking, including over-the counter medications, herbal remedies, vitamins, and supplements.
* The patient will be asked about any disease-related symptoms they are experiencing.
* The patient will receive a new supply and the medication diary will be reviewed.

Every 12 weeks (+/-1 week) the following procedures will be performed in clinic:

* Blood tests. A small sample of the patient's blood (about 1-2 tablespoons) will be collected. This blood will be collected for specialized laboratory tests.
* A (CT) scan of the patient's chest and a CT or MRI scan of abdomen, and pelvis and a bone scan will be performed every 12 weeks (+/- 1 week) while the patient is on active treatment. If your baseline CT of the patient's chest does not show disease, the investigator may not asked for this to be repeated.

End of Study Visit in clinic:

* A medical history.
* A physical examination
* Performance status
* Blood tests (2-3 tablespoons)
* The patient will be asked about any disease-related symptoms If the patient completed at least 4 cycles of enzalutamide, the patient will undergo a second of two required biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Be a male ≥ 18 years of age.
* Participants must have histologically or cytologically confirmed adenocarcinoma of the prostate without ≥50% neuroendocrine differentiation or small cell histology.
* Participants must have progressive disease as defined by either:
* Castrate resistant disease as defined by PCWG. Participants must have a rise in PSA on two successive determinations at least one week apart and PSA levels ≥ 2 ng/ml (only the screening PSA needs to be ≥ 2 ng/ml) and testosterone levels < 50 ng/dL, OR
* Soft tissue progression defined by RECIST 1.1, OR
* Bone disease progression defined by PCWG2 with two or more new lesions on bone scan.
* CRPC with metastatic disease with at least one site of metastatic disease must be amenable to needle biopsy. Soft tissue biopsy sites include: lymph node or visceral metastases. Bone sites include lumbar vertebrae, pelvic bones and long bones. Excluded sites are thoracic, cervical vertebrae, skull and rib lesions. Biopsy site will be selected with guidance of interventional radiologist determining best site to optimize balance of obtaining useful tissue for analysis and minimizing risk.
* Participants without orchiectomy must be maintained on LHRH agonist/antagonist therapy.
* Participants may have had any number of previous hormonal therapies (antiandrogens, steroids, estrogens, finasteride, dutasteride, ketoconazole, abiraterone) provided these were discontinued ≥ 4 weeks before enrollment.
* Participants may have had up to two previous cytotoxic therapeutic regimens provided these were discontinued ≥ 4 weeks before enrollment.
* At least a 4 week interval from previous prostate cancer treatment other than LHRH agonist/antagonist therapy or bisphosphonates to enrollment.
* Participants receiving bisphosphonates therapy can be maintained on this therapy. If participants have not started bisphosphonates, it is recommended that they start treatment after the first biopsy.
* ECOG performance status < 2 (Karnofsky >60%, see Appendix A).
* Participants must have normal organ and marrow function as defined below:
* WBC ≥ 3,000/mcL
* ANC ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Hemoglobin ≥ 9 g/dL
* Serum albumin ≥ 3.0 g/dL
* AST, ALT, and total bilirubin ≤ 1.5 x Institutional ULN
* Creatinine ≤ 1.5 Institutional ULN or a calculated creatinine clearance ≥ 50 mL/min using the Cockcroft Gault equation
* PTT ≤ 60, INR ≤ 1.5 Institutional ULN unless on warfarin therapy (investigator would need to determine if safe for participant to stop warfarin prior to biopsy)
* Have signed an informed consent document indicating that the subjects understands the purpose of and procedures required for the study and are willing to participate in the study.
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol.
* Written Authorization for Use and Release of Health and Research Study Information (US sites only) has been obtained.
* Able to swallow the study drug whole as a tablet.
* Participants who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator during the treatment period and for 1 week after last dose of enzalutamide.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements within 6 months of enrollment.

Clinically significant heart disease as evidenced by:

* Myocardial infarction within 6 months of enrollment.
* Uncontrolled angina within 6 months of enrollment.
* Congestive heart failure NYHA Class III or IV, or a history of congestive heart failure NYHA Class III or IV in the past, unless a screening ECHO or MUGA within 3 months results in a left ventricular ejection fraction ≥ 45%.
* Clinically significant ventricular arrhythmias.
* History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place.
* Bradycardia as indicated by a heart rate < 50 beats per minute at screening visit.
* Hypotension as indicated by SBP ≤ 85 on 2 consecutive measurements.
* Uncontrolled hypertension as indicated by SBP > 170 mmHg or DBP > 105 mmHg on 2 consecutive measurements at screening visit.
* Thromboembolism within 6 months of enrollment.
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
* History of seizure or any condition or concurrent medication that may predispose to seizure.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances: 1) individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy, or 2) individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: superficial bladder cancer, basal cell or squamous cell carcinoma of the skin.
* Known brain metastasis. Participants with brain metastasis can only be included if they were treated > 4 week prior to enrollment with radiation and the effects of treatment have resolved. Subjects with treated brain metastases must have a post-treatment brain MRI showing no further progression of prior lesions and no new metastatic lesions. Subjects will be ineligible if they have any ongoing symptoms from brain metastases or if there continues to be radiographic evidence of cerebral edema.
* Have known allergies, hypersensitivity, or intolerance to enzalutamide or their excipients.
* Surgery or local prostatic intervention within 30 days of the first dose. In addition, any clinically relevant issues from the surgery must have resolved prior to enrollment.
* Major surgery or radiation therapy within 4 weeks of enrollment. Radium-223, strontium-89, or samarium-153 therapy within 4 weeks of enrollment. Radiotherapy, chemotherapy or immunotherapy within 4 weeks, or single fraction of palliative radiotherapy within 14 days of administration of enrollment.
* Prior treatment with enzalutamide.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of enrollment.
* Concomitant use of medications that may alter pharmacokinetics of enzalutamide. See section 5.3.
* Any acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a NCI CTCAE (version 4) grade of ≤ 1. Chemotherapy induced alopecia and grade 2 peripheral neuropathy are allowed.
* Condition or situation which, in the investigator's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with participant's participation in the study.
* Individuals not willing to comply with the procedural requirements of this protocol.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with enzalutamide. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-09-13 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - University of Washington Medical Center/Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sperger JM, Emamekhoo H, McKay RR, Stahlfeld CN, Singh A, Chen XE, Kwak L, Gilsdorf CS, Wolfe SK, Wei XX, Silver R, Zhang Z, Morris MJ, Bubley G, Feng FY, Scher HI, Rathkopf D, Dehm SM, Choueiri TK, Halabi S, Armstrong AJ, Wyatt AW, Taplin ME, Zhao SG, Lang JM. Prospective Evaluation of Clinical Outcomes Using a Multiplex Liquid Biopsy Targeting Diverse Resistance Mechanisms in Metastatic Prostate Cancer. J Clin Oncol. 2021 Sep 10;39(26):2926-2937. doi: 10.1200/JCO.21.00169. Epub 2021 Jul 1. PMID 34197212

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide: Participants will be treated with four 40 mg capsules (160 mg) once daily of enzalutamide taken orally with 28-days cycle. Participants will maintain a drug diary from time of initiation of study treatment to time of discontinuation from the study (Appendix C).
Period: Overall Study
Arm/Group | Enzalutamide
Started | 67
Completed | 0
Not Completed | 67
Not completed — Death | 1
Not completed — Symptomatic or radiographic progression | 49
Not completed — Adverse Event | 6
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2
Not completed — Intercurrent Illness | 1
Not completed — On treatment | 3
Not completed — Never initiate the treatment | 2

BASELINE CHARACTERISTICS:
Population: Patients who received ≥1 dose of enzalutamide. Two patients didn't initiate the treatment.
Groups:
- Enzalutamide: Participants will be treated with four 40 mg capsules (160 mg) once daily of enzalutamide taken orally. All participants without orchiectomy will be maintained on LHRH agonist/antagonist therapy. Participants will be evaluated clinically and with laboratory studies on day 1 of every 28 day cycle. Participants will maintain a drug diary from time of initiation of study treatment to time of discontinuation from the study (Appendix C).
  Enzalutamide: Administration: 160 mg orally once daily. Treatment will be continued until evidence of symptomatic or radiographic progression or the participant is taken off the study for another reason.
  Dosing: 160 mg orally taken once daily as four 40 mg capsules.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 65
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [66 to 75]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 51
  More than one race | 1
  Unknown or Not Reported | 8
Institution [Count of Participants; unit: Participants]
  Dana-Farber Cancer Institute | 39
  University of Washington | 19
  Beth Israel Deaconess Medical Center | 6
  South Shore Hospital | 1
Prior chemotherapy [Count of Participants; unit: Participants]
  Yes | 16
  No | 49
Prior docetaxel [Count of Participants; unit: Participants]
  Yes | 15
  No | 50
Prior abiraterone [Count of Participants; unit: Participants]
  Yes | 22
  No | 43
Prior ketoconazole [Count of Participants; unit: Participants]
  Yes | 9
  No | 56

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Gene Alterations
Description: Serial biopsies was performed at pre-study and progression to analyze mechanisms of resistance to enzalutamide, such as alterations in AR (mutations, amplifications), tumor suppression genes, DNA repair genes, and SPOP. Whole exome sequencing was performed on tumor tissue biopsies.
Time Frame: Tumor biopsies were performed at pre-study and progression. Progression occurred up to 41 months after initiation of enzalutamide.
Population: Patients who had paired biopsies of pre-study and progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 10
Participants
  AR amplifications at pre-study | 7
  AR mutations at pre-study | 4
  TP53 alteration at pre-study | 7
  RB1 alteration at pre-study | 7
  PTEN alteration at pre-study | 6
  BRCA2 alteration at pre-study | 4
  CDK12 alteration at pre-study | 1
  ATM alteration at pre-study | 1
  SPOP alteration at pre-study | 4

2. Secondary Outcome: Changes in Serum Androgen Concentrations Between Baseline and Subsequent Assessment Visits
Description: Serum testosterone were be collected at pre-study (C1D1) and every cycle and changes over time from baseline were planned to be summarized descriptively.
Time Frame: Not collected.
Population: Serum data on the trial was collected but hormone assays were not run due to insufficient funding.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With a PSA Response
Description: PSA response is defined per PCWG2 criteria (PSA decline >=50% relative to cycle 1 PSA) and is summarized as frequency and percent.
Time Frame: PSA was measured at pre-treatment, each C1D1 (1 cycle=28 days), end of treatment, and follow-up visits (every 6 months). PSA were measured up to 52 months.
Population: Patients who received ≥1 dose of enzalutamide
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 65
Participants
  ≥50% PSA reduction | 38
  ≥90% PSA reduction | 20

4. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response is defined as time from the first achievement of PSA response (PSA decline >=50% from cycle 1) to the date of PSA progression or death, whichever occurs first.
Time Frame: as for outcome 3
Population: Patients who experienced PSA response defined as more than equal to 50% decline from baseline.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 38
months | 3.2 [1.4 to 7.4]

5. Secondary Outcome: Response of Measurable Disease at Baseline
Description: Objective responses for measurable disease was evaluated using RECIST 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Response was tabulated with frequency.
Time Frame: Imaging was performed at pre-study and every 12 weeks on treatment. Treatment cycles is 28 days. Patients were assessed up to 41 months.
Population: Patients with measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 32
Participants
  Complete response | 0
  Partial response | 11
  Stable disease | 11
  Progressive disease | 7
  Inevaluable/missing | 3

6. Secondary Outcome: Duration of Response of Measurable Disease
Description: Duration of response of measurable disease is defined as time from the date of first objective response (PR/CR) to date of progression or death, whichever comes first.
  Objective response is per RECIST 1.1 criteria:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 5
Population: Patients with CR or PR to enzalutamide. There was no CR achieved and 11 PRs.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Enzalutamide
Number analyzed (Participants) | 11
months | 2.8 [0.03 to 7.8]

7. Secondary Outcome: Toxicity Measurements
Description: For safety and tolerability, treatment-related grade 3 or higher toxicities was assessed using CTCAE v. 4.0 and was provided using frequency.
Time Frame: Toxicity was reported at pre-study, every cycle, and end of treatment visit. Patients reported toxicities up to 39 months.
Population: Patients who received at least one dose of enzalutamide.
Measure: Count of Participants; unit: Participants
Groups:
- Enzalutamide: Participants will be treated with four 40 mg capsules (160 mg) once daily of enzalutamide taken orally with 28-days cycle. Participants will maintain a drug diary from time of initiation of study treatment to time of discontinuation from the study (Appendix C).
  Enzalutamide: Administration: 160 mg orally once daily. Treatment will be continued until evidence of symptomatic or radiographic progression or the participant is taken off the study for another reason.
  Dosing: 160 mg orally taken once daily as four 40 mg capsules.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 65
Participants
  Grade 3 hypertension | 4
  Grade 3 colitis | 1
  Grade 3 fatigue | 1

8. Secondary Outcome: Number of Participants With PSA Response Stratified by Gene Alterations in Serial Tumor Biopsies
Description: Serial biopsies was performed at pre-study and progression to analyze mechanisms of resistance to enzalutamide, such as alterations in AR (mutations, amplifications), DNA repair genes, and SPOP. Whole exome sequencing was performed on tumor tissue biopsies. Gene alterations were tabulated with PSA response.
Time Frame: Tumor biopsies will be performed at pre-treatment and end of treatment visit. Treatment cycle is 28 days. PSA was collected up to 52 months.
Population: Patients who had paired biopsies of pre-study and progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 10
Participants
  PSA response among patients in Patients with AR amplification | 3
  PSA response among patients with AR mutation | 1
  PSA response among patients with SPOP alteration | 2

9. Secondary Outcome: Subsequent Lines of Therapy
Description: Subsequent lines of therapy following study drug discontinuation was summarized descriptively.
Time Frame: Subsequent treatments were followed up to 31 months after discontinuation of study drug.
Population: Patients who received at least one dose of enzalutamide.
Measure: Median (Inter-Quartile Range); unit: Lines of treatment
Arm/Group | Enzalutamide
Number analyzed (Participants) | 65
Lines of treatment | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: Toxicities were assessed every cycle and up to 30 days after coming off from the treatment. Toxicities were collected up to ~ 44 months.
Description: A serious adverse event (SAE) is any adverse event, occurring at any dose and regardless of causality that:
  * Results in death
  * Is life-threatening. Life-threatening means that the person was at immediate risk of death from the reaction as it occurred, i.e., it does not include a reaction which hypothetically might have caused death had it occurred in a more severe form.
  * Requires or prolongs inpatient hospitalization
  * Results in persistent or significant disability/incapacity
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 41/65
Serious Adverse Events (participants affected / at risk) | 8/65
Other Adverse Events (participants affected / at risk) | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=65)
Cardiac arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=65)
Anemia (Blood and lymphatic system disorders) | 11
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrioventricular block first degree (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 3
Vertigo (Ear and labyrinth disorders) | 4
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 1
Eye pain (Eye disorders) | 1
Floaters (Eye disorders) | 1
Retinal vascular disorder (Eye disorders) | 1
Watering eyes (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 5
Abdominal pain (Gastrointestinal disorders) | 3
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophageal obstruction (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Oral pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema limbs (General disorders) | 7
Fatigue (General disorders) | 34
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
Irritability (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 23
General disorders and administration site conditions - Other, specify (General disorders) | 2
Bronchial infection (Infections and infestations) | 3
Eye infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 3
Infections and infestations - Other, specify (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 6
Fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 20
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 11
Dysesthesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 4
Encephalopathy (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 4
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 6
Libido decreased (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 1
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 5
Renal calculi (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 8
Urinary incontinence (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3
Breast pain (Reproductive system and breast disorders) | 4
Erectile dysfunction (Reproductive system and breast disorders) | 2
Genital edema (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 5
Pelvic pain (Reproductive system and breast disorders) | 4
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4
Flushing (Vascular disorders) | 2
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 20
Hypertension (Vascular disorders) | 18
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT01942837/Prot_SAP_000.pdf